CLINICAL TRIAL: NCT05297513
Title: Efficacy of ActiveMatrix on Spinal Surgical Site Infection (SSI) Reduction: A Single-blinded Randomized Controlled Trial
Brief Title: Efficacy of ActiveMatrix on Spinal SSI Rate
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Skye Biologics Holdings, LLC (Industry)
Responsible Party: Principal Investigator, Alfonso Fuentes, MD, Assistant Professor Neurosurgery BCM, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-51093
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Spinal Stenosis Lumbar; Surgical Site Infection; Back Pain Lower Back Chronic
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment, no intervention (No Intervention)
- Standard treatment, plus ActiveMatrix (Experimental)
  Interventions: Drug: ActiveMatrix

INTERVENTIONS:
Drug: ActiveMatrix — All patients will receive weight based prophylactic antibiotics i.e. Ancef, vancomycin, or clindamycin. Drains will be used in fusion cases only. Intrawound vancomycin will be used for all instrumented cases.No negative pressure devices will be used. Anatomic layers will be closed in similar, standard fashion for all cases. For those randomized to the treatment group, the ActiveMatrix product will be administered on top of the dura mater and again on the closed fascia. Those in the control group, will forgo this step.
  Arms: Standard treatment, plus ActiveMatrix

SUMMARY:
This clinical trial seeks to provide high level of evidence on the efficacy of ActiveMatrix primarily on spinal surgical site infection rate.

DETAILED DESCRIPTION:
Postoperative spinal surgical site infections (SSI) have a significant effect on patient morbidity and mortality.1 Spinal SSI as well as other complications including pseudoarthrosis occur at a higher rate in patients with comorbidities including obesity, smoking history, diabetes, steroid use, older age, and higher modified frailty index.2 Patients of Veterans Affairs (VA) medical centers have higher number of comorbidities than non-VA patients, and are therefore at higher risk for postoperative spinal SSI and complications.3,4 Spinal SSI has been reported to be anywhere from <1% in decompressions to >10% after instrumented fusion.5 Anecdotal evidence has suggested SSI to be as high as 20% among our population. As spine surgeons for the largest VA in the country, our team sought a product that could reduce the rate of spinal SSI, and ideally result in improved patient outcomes, in our at-risk patient population.

Skye Biologics offers placental tissue-based matrices in the form of both flowable and solid mediums. The flowable matrix has been shown in-vitro to contain significant amounts of collagen and growth factors, as well as molecules known to modulate immune response. The results of this have been in-vitro inhibition of methicillin resistant Staphylococcus aureus (MRSA) and Staphylococcus saprophyticus proliferation, increase in migration of adipose-derived stem cells (ASCs), adherence to the ASCs in cultures.6 In translation of these results clinical application has been well received, with various subspecialties including ENT and orthopedics using the products. Based on both the positive in vitro and in vivo results, out team began using the flowable product with good initial subjective results, including improved wound healing and excellent patient satisfaction. The true clinical efficacy remains to be assessed, however. Our team sought to provide level 1 evidence on this product in thoracolumbosacaral posterior spinal decompression and/or fusion in our at-risk population via a single-blinded randomized control trial at high-volume institution (s).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ≥ 18 years of age to 100 years of age
4. Have a clinical diagnosis of thoracic and or lumbosacral spinal disease indicated for decompression and/or fusion
5. Have no contraindications or allergies to the treatment administered

Exclusion Criteria:

1. Subject is involved with a worker's compensation, personal injury, or other legal matters related to their health
2. Subject does not provide full consent
3. Known history of allergy to allografts
4. Pregnancy or lactation
5. Minimally invasive spinal surgery
6. Non-fusion instrumented cases requiring drains

There is no intended distribution or restriction of subjects by racial and ethnic origin. No vulnerable subjects are included in this protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
90-day surgical site infection | 90 days

SECONDARY OUTCOMES:
Fascial defects at 3-6 months for fusion cases | 6 months
Improvement in back and leg pain | 6 months
  Oswestry Low Back Disability Questionnaire/Index (0-100, higher scores indicate greater disability)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casper DS, Zmistowski B, Hollern DA, Hilibrand AS, Vaccaro AR, Schroeder GD, Kepler CK. The Effect of Postoperative Spinal Infections on Patient Mortality. Spine (Phila Pa 1976). 2018 Feb 1;43(3):223-227. doi: 10.1097/BRS.0000000000002277. PMID 28604484
- [Background] Badiee RK, Mayer R, Pennicooke B, Chou D, Mummaneni PV, Tan LA. Complications following posterior cervical decompression and fusion: a review of incidence, risk factors, and prevention strategies. J Spine Surg. 2020 Mar;6(1):323-333. doi: 10.21037/jss.2019.11.01. PMID 32309669
- [Background] Melzer AC, Pinsker EA, Clothier B, Noorbaloochi S, Burgess DJ, Danan ER, Fu SS. Validating the use of veterans affairs tobacco health factors for assessing change in smoking status: accuracy, availability, and approach. BMC Med Res Methodol. 2018 May 11;18(1):39. doi: 10.1186/s12874-018-0501-2. PMID 29751746
- [Background] Agha Z, Lofgren RP, VanRuiswyk JV, Layde PM. Are patients at Veterans Affairs medical centers sicker? A comparative analysis of health status and medical resource use. Arch Intern Med. 2000 Nov 27;160(21):3252-7. doi: 10.1001/archinte.160.21.3252. PMID 11088086
- [Background] O'Toole JE, Eichholz KM, Fessler RG. Surgical site infection rates after minimally invasive spinal surgery. J Neurosurg Spine. 2009 Oct;11(4):471-6. doi: 10.3171/2009.5.SPINE08633. PMID 19929344
- [Background] Irvin J, Danchik C, Rall J, Babcock A, Pine M, Barnaby D, Pathakamuri J, Kuebler D. Bioactivity and composition of a preserved connective tissue matrix derived from human placental tissue. J Biomed Mater Res B Appl Biomater. 2018 Nov;106(8):2731-2740. doi: 10.1002/jbm.b.34054. Epub 2018 Feb 13. PMID 29437272
- See also: Related Info — https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf.